CLINICAL TRIAL: NCT04277312
Title: Project Daire: Derry/Londonderry as the Nexus City for Food, Education, Trust and Health'
Brief Title: Project Daire: Derry/Londonderry as the Nexus City for Food, Education, Trust and Health
Acronym: Daire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Invest NI (Unknown)
Responsible Party: Principal Investigator, Jayne Woodside, PhD, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 038_1819; RD1014267 (Other Grant/Funding Number: Invest NI)
Record Dates: First submitted 2020-02-11; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: Primary School Children; Food Education; Food Knowledge; Childhood Health; Childhood Wellbeing
MeSH Terms: conditions — Behavior | interventions — engage 8200

STUDY DESIGN:
Intervention Model Description: Project Daire is a randomised-controlled, factorial design trial evaluating two interventions
Masking Description: Masking was not possible due to the nature of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Engage (Experimental): The Engage intervention was developed with input from primary school teachers and includes a range of age-appropriate educational activities related to food. Activities include videos, lesson plans, worksheets, games, talks/visits from experts, visits to industrial partners and other local food-related centres of interest and practical activities such as experiments. All 'Engage' material is mapped to the Northern Ireland School Curriculum. The 'Engage' intervention is structured into three broad topics: Farm to Fork; Pleasure on a Plate and Food Futures. Engage resources were provided to schools electronically and in hard copy and teachers delivered most of the content, with the exception of several sessions which were delivered by visiting scientists.
  Interventions: Behavioral: Engage
- Nourish (Experimental): The Nourish intervention is a school food environment intervention which included weekly healthy snack provision supplied by food industry partners, enhancement of canteen dining area (café style, tablecloths, centre pieces, bunting and menu boards, healthy eating posters), attendance at Tasting Days held in Higher Education Colleges (children were encouraged to try new foods provided by industry partners and received stamps on 'food passports' in return) and sensory educational and cookery activities.
  Interventions: Behavioral: Nourish
- Nourish and Engage (Experimental): This arm of the intervention delivered both the Nourish and Engage interventions as detailed above.
  Interventions: Behavioral: Engage; Behavioral: Nourish
- Delayed (No Intervention): The delayed arm of the intervention was the control arm. Schools randomised to this arm of the study were offered the Engage intervention resources after endpoint data collection.

INTERVENTIONS:
Behavioral: Engage — The Engage intervention was developed with input from primary school teachers and includes a range of age-appropriate educational activities related to food. Activities include videos, lesson plans, worksheets, games, talks/visits from experts, visits to industrial partners and other local food-related centres of interest and practical activities such as experiments. All 'Engage' material is mapped to the Northern Ireland School Curriculum. The 'Engage' intervention is structured into three broad topics: Farm to Fork; Pleasure on a Plate and Food Futures. Engage resources were provided to schools electronically and in hard copy and teachers delivered most of the content, with the exception of several sessions which were delivered by visiting scientists.
  Arms: Engage; Nourish and Engage
Behavioral: Nourish — The Nourish intervention is a school food environment intervention which included weekly healthy snack provision supplied by food industry partners, enhancement of canteen dining area (café style, tablecloths, centre pieces, bunting and menu boards, healthy eating posters), attendance at Tasting Days held in Higher Education Colleges (children were encouraged to try new foods provided by industry partners and received stamps on 'food passports' in return) and sensory educational and cookery activities.
  Arms: Nourish; Nourish and Engage

SUMMARY:
Project Daire is a randomised-controlled factorial design trial working in partnership with primary schools and local food producers evaluating two interventions designed to improve primary school children's knowledge of and interest in food and where it comes from, with the ultimate aim of driving improvement in health, well-being and educational status.

DETAILED DESCRIPTION:
Project Daire is a randomised-controlled factorial design trial working in partnership with primary schools and local food producers evaluating two interventions designed to improve primary school children's knowledge of and interest in food and where it comes from, with the ultimate aim of driving improvement in health, well-being and educational status. Key Stage 1 and 2 pupils will be recruited from 15 primary schools in the North West of Northern Ireland and will be randomised to one of four intervention arms: i) 'Engage', ii) 'Nourish', iii) 'Engage' and 'Nourish' and iv) Delayed of duration up to 6 months. Study outcomes include food knowledge, attitudes, trust, diet, behaviour, health and wellbeing and will be collected at baseline and six months.

ELIGIBILITY:
Inclusion Criteria:

* Mainstream primary schools willing to be randomly assigned to an intervention,
* Mainstream primary schools willing to engage with the intervention and implement it with their pupils,
* Mainstream primary schools willing to facilitate pre and post-test data collection in their setting,
* Mainstream primary schools within the North West region of Northern Ireland.
* Pupils in Primary 3 (Key Stage 1) and Primary 7 (Key Stage 2) of participating schools were eligible to take part.

Exclusion criteria

* Secondary schools
* Non-mainstream schools
* Schools not in the North West region of Northern Ireland

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1080 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Change in KIDSCREEN-10 score at 6 months | Baseline (Month 0), 6 months
  Validated well-being questionnaire for children. Completed by KS1 and KS2 pupils.This is an 11-item instrument answered on a 5-point scale and results in one global HRQoL score. Most of the items are formulated positively and in concordance with the scoring, which means a higher score reflects a higher HRQoL. However, some items are formulated negatively and as a consequence the scoring has to be recoded. The scoring method results in T-values with scale means around 50 and standard deviations around 10 with higher values indicating higher HRQoL.
Change in Strengths and Difficulties Questionnaire score at 6 months | Baseline (Month 0), 6 months
  Validated brief behavioural screening questionnaire. Completed by teachers. This 25-item instrument incorporates 5 scales of 5 items, with each item answered on a 3 point scale. All scales represent a negative trait, with the exception of the ProSocial Scale which indicates a positive trait. For each of the 5 scales the score can range from 0 to 10 if all items were completed. A Total Difficulties score is the final score and indicates poorer behaviour. Therefore the lower the score, the better the outcome in terms of behaviour.

SECONDARY OUTCOMES:
24 Hour Dietary Record | Baseline (Month 0), 6 months
  Validated dietary intake questionnaire in age group (Moore et al., Br J Nutr 2008;99:1266-74). Completed by KS1 and KS2 pupils. Prospective record of all foods and drinks consumed over a 24 hour period. Data are analysed using dietary analysis software to produce average daily intake of food groups, macronutrients, micronutrients, vitamins and minerals.
Food Frequency Questionnaire | Baseline (Month 0), 6 months
  Food Frequency Questionnaire developed by study team based on other similar age-appropriate food frequency questionnaires (Cade et al., Public Health Nutr 2005;9:501-8). Two versions-one shorter version developed for younger KS1 age group, one for KS2 age group. Children asked to indicate categorical responses ('yes', 'no' and 'not sure') to indicate whether or not they ever eat a particular food. Presented as a food group list with categorical responses.
Food Shopping, Preparation & Consumption | Baseline (Month 0), 6 months
  Questionnaire developed by study team. Completed by KS1 and KS2 pupils. Children asked to indicate categorical responses 'always', 'sometimes', 'never' or 'agree' 'not sure' or 'do not agree' with reference to various cooking, food preparation scenarios and how they feel about trying new foods.
Perceived cooking competence | Baseline (Month 0), 6 months
  Researcher developed questionnaire (items sourced from unpublished data), based on similar measures for perceived movement competence (Barnett et al., 2015; Harter and Pike, 1984). Completed by KS1 and KS2 pupils-shorter version developed for KS2 pupils. Categorical responses 'yes' and 'no' with regards to have they ever demonstrated a range of different cooking skills. Children are then presented with a range of illustrated characters who vary in their competence and child indicates which child they are most like with regards to that particular cooking skill.
Agri-Food Knowledge | Baseline (Month 0), 6 months
  Questionnaire designed to assess pupil knowledge on range of agri-food topics (food chain, farm, seasonality, local versus imported). Researcher developed with industry input, piloted and face validity with experts in the different fields, some items adapted from previous measures (Moss et al., 2013; Reynolds et al., 2012; Harmon and Maretzki, 2006; Saksvig et al., 2005) and BNF - Food a fact of Life (http://archive.foodafactoflife.org.uk/Activity.aspx?siteId=14&sectionId=63&contentId=176). Completed by KS1 and KS2 pupils-shorter version developed for KS1 pupils. Responses categorical and categories varied by item type.
Food Jobs/Careers Aspirations | Baseline (Month 0), 6 months
  Questionnaire to assess career aspirations and knowledge of food-related jobs. Developed by research team. Completed by KS1 and KS2 pupils. Open-ended questions asking about career aspirations and assessing knowledge of careers related to food.
Preference/Willingness to Try | Baseline (Month 0), 6 months
  Questionnaire to assess knowledge of willingness to try range of foods. Researcher adapted from Morgan et al. (2010) and Birch and Sullivan (1991). Completed by KS1 and KS2 pupils-shorter version for KS1 pupils.Responses largely categorical with some open-ended questions asking children to identify the food.
Attitudes | Baseline (Month 0), 6 months
  Questionnaire to assess pupil attitude to importance of health behaviours, including diet. Previously used in a survey of NI schoolchildren health (Young Hearts Studies). Completed by KS2 pupils only. This is an 11-item instrument assessing attitudes towards importance of various health behaviours 'very important', 'quite important', 'not important'
Food source to product - knowledge | Baseline (Month 0), 6 months
  Questionnaire to assess level of knowledge in terms of food source to product. Developed by research team. Completed by KS1 and KS2 pupils. Categorical matching responses.
Trust | Baseline (Month 0), 6 months
  Questionnaire to assess level of trust in local food products. Developed by research team. Completed by KS2 only. This is a 10-item instrument answered on a 5-point scale (definitely disagree, disagree, not sure, agree, definitely agree).
School food environment observation | Baseline (Month 0), 6 months
  Observational proforma designed to allow researcher to assess current school food environment. Developed by research team. Completed by researcher. Observational-open-ended responses.
School food environment questionnaire | Baseline (Month 0), 6 months
  Questionnaire designed to assess current school food environment. Developed by research team. Completed by school principal/management
Exposure to/Experience with Agri-Food | Baseline only (Month 0)
  Questionnaire designed to characterise pupils in terms of previous experience of agri-food. Developed by research team. Developed with KS1 and KS2 age-appropriate questions. Categorical responses.
Baseline Skills Scale | Baseline only (Month 0)
  Questionnaire designed to characterise pupil's level of cooking skills. Previously validated questionnaire. Children indicate how good they believe they are at various cooking skills on a 7-point scale (1 is very poor and 7 is very good).
Daire Evaluation questionnaire | 6 months only
  Process Evaluation questionnaire for both Nourish and Engage interventions completed by teachers. Developed by research team. Categorical and op-ended responses.

CONTACTS AND LOCATIONS:
Overall Officials: Jayne Woodside, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Centre for Public Health, Queen's University Belfast, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anderson N, Brennan SF, Lavelle F, Moore SE, Olgacher D, Junkin A, Dean M, McKinley MC, McCole P, Hunter RF, Dunne L, O'Connell NE, Elliott CT, McCarthy D, Woodside JV. Process evaluation of Project Daire: a food environment intervention that impacted food knowledge, wellbeing and dietary habits of primary school children. BMC Public Health. 2025 Feb 6;25(1):486. doi: 10.1186/s12889-025-21628-4. PMID 39910503
- [Derived] Brennan SF, Lavelle F, Moore SE, Dean M, McKinley MC, McCole P, Hunter RF, Dunne L, O'Connell NE, Cardwell CR, Elliott CT, McCarthy D, Woodside JV. Food environment intervention improves food knowledge, wellbeing and dietary habits in primary school children: Project Daire, a randomised-controlled, factorial design cluster trial. Int J Behav Nutr Phys Act. 2021 Feb 4;18(1):23. doi: 10.1186/s12966-021-01086-y. PMID 33541372